CLINICAL TRIAL: NCT03229707
Title: Impact Of Digital Photography & Conventional Method On The Accuracy Of Shade Matching In The Esthetic Zone
Brief Title: Impact Of Digital Photography & Conventional Method On The Accuracy Of Dental Shade Matching In The Esthetic Zone
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Rawan Ferroukhi, Master Student, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Screening
Other Study IDs: CEBC-CU-2017-07-17
Record Dates: First submitted 2017-07-23; First posted 2017-07-25 (Actual); Last update posted 2021-07-29 (Actual); Status verified 2021-07

CONDITIONS: Accuracy of Dental Shade Selection in the Aesthetic Zone

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group 1 Color matching using Vita 3D master (Active Comparator): Outcome Name: Color Matching measured by :
  Modified (USPHS) criteria
  Interventions: Device: Vita 3D master shade guide
- group 2 Color matching using digital photography (Experimental): Outcome Name: Color Matching measured by Digital Photography using (Photoshop)
  Software:
  * 0 to 1: no difference in perception
  * 1 to 2: only perceptible to a trained observer
  * 2 to 3.5: perceptible difference
  * 3.5 to 5: marked difference
  Interventions: Device: Digital photography using software Photoshop

INTERVENTIONS:
Device: Digital photography using software Photoshop — When taking the image, a gray card is used for subsequent exposure calibration in Adobe Camera Raw (which is packaged with Photoshop).
  * Images are then opened into Photoshop.
  * The "INFO" panel must be open.
  * Click on the small eyedropper in the Info panel window and click on ''Lab Color".
  * Place the mouse over the center of the tooth to be measured for L value.
  * Click on the "HSB Color" option, which stands for hue, saturation, and brightness.
  Arms: group 2 Color matching using digital photography
Device: Vita 3D master shade guide — Alpha (A)Perfectly matched Beta (B)Not perfectly matched Charlie (C)unacceptable Determent by 10 observers
  Other Names: Conventional shade matching
  Arms: group 1 Color matching using Vita 3D master

SUMMARY:
The aim of this study:

Is to evaluate the accuracy of digital photography in optimizing shade matching when compared to conventional method of shade selection.

DETAILED DESCRIPTION:
Randomized control trial, 2 groups will be included. Group 1: Color matching using Vita 3D master, using modified (USPHS) criteria Group 2: Color matching using digital photography using (Photoshop adopt) the assessment will be through a questionnaire for the patient satisfaction outcome using Visual analogue scale

ELIGIBILITY:
Inclusion Criteria:

1. Patients between 18-70 years old, able to read and sign the informed consent document.
2. Patients requiring restorations in the esthetic zone.
3. Patients don't have active periodontal or pulpal diseases
4. Patients willing to return for follow-up examination and evaluation.

Exclusion Criteria:

1. Patients in the growth stage.
2. Patients with poor oral hygiene and lack of motivation.
3. Psychiatric problems or unrealistic expectations.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2018-07-01 (Actual); Primary Completion 2018-10-31 (Actual); Study Completion 2019-08-01 (Actual)

PRIMARY OUTCOMES:
Patient satisfaction | 1 year
  Visual analogue scale

SECONDARY OUTCOMES:
Color Matching | 1 year
  Digital Photography using (Photoshop)/using Vita 3D master Modified (USPHS) criteria

CONTACTS AND LOCATIONS:
Overall Officials: Rawan Ferroukhi, Masters in FixedProsthodontics, Principal Investigator — MSc Student of Fixed Prosthodontics, Division of Fixed Prosthodontics, Faculty of Dentistry, Cairo University, Cairo, Egypt
Locations (1):
- Cairo University, Cairo, Egypt

REFERENCES:
- See also: Related Info — https://www.actascientific.com/ASDS/pdf/ASDS-04-0945.pdf